CLINICAL TRIAL: NCT05590403
Title: A Phase 3, Observer-blind, Randomized, Placebo-controlled Study to Evaluate the Non-inferiority of the Immune Response and Safety of the RSVPreF3 OA Investigational Vaccine in Adults 50-59 Years of Age, Including Adults at Increased Risk of Respiratory Syncytial Virus Lower Respiratory Tract Disease, Compared to Older Adults ≥60 Years of Age
Brief Title: A Study on the Immune Response and Safety of a Vaccine Against Respiratory Syncytial Virus Given to Adults 50-59 Years of Age, Including Adults at Increased Risk of Respiratory Syncytial Virus Lower Respiratory Tract Disease, Compared to Older Adults 60 Years of Age and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 219238; 2022-001981-36 (EudraCT Number)
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Immunogenicity; Safety; Increased risk of respiratory syncytial virus lower respiratory tract disease; Adults aged 50-59 years of age; Older adults 60 years of age and above
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind for Cohort 1 (Day1-Day 31) and single-blind afterwards and open-label for Cohort 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Adults HA-RSV Group (Experimental): Healthy adults or adults with chronic stable conditions with or without treatment that do not lead to an increased risk of RSV-Lower respiratory tract disease (RSV-LRTD), aged 50-59 years old received 1 dose of RSVPreF3 OA vaccine at Day 1 and were followed until study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Adults HA-Placebo Group (Placebo Comparator): Healthy adults or adults with chronic stable conditions with or without treatment that do not lead to an increased risk of RSV-LRTD, aged 50-59 years old received 1 dose of placebo at Day 1 and were followed until study end.
  Interventions: Drug: Placebo
- Adults AIR-RSV Group (Experimental): Adults at increased risk of RSV-Lower respiratory tract disease (RSV-LRTD) aged 50-59 years old received 1 dose of RSVPreF3 OA vaccine at Day 1 and were followed until study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- Adults AIR-Placebo Group (Placebo Comparator): Adults at increased risk of RSV-LRTD aged 50-59 years old received 1 dose of placebo at Day 1 and were followed until study end.
  Interventions: Drug: Placebo
- OA-RSV Group (Experimental): Older adults aged 60 years old and above received 1 dose of RSVPreF3 OA vaccine at Day 1 and were followed until study end.
  Interventions: Biological: RSVPreF3 OA investigational vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — One dose administered intramuscularly at Day 1.
  Arms: Adults AIR-RSV Group; Adults HA-RSV Group; OA-RSV Group
Drug: Placebo — One dose administered intramuscularly at Day 1.
  Arms: Adults AIR-Placebo Group; Adults HA-Placebo Group

SUMMARY:
The aim of this study is to demonstrate the non-inferiority (NI) of the immune response and evaluate safety of RSVPreF3 older adults (OA) investigational vaccine in adults 50-59 years of age (YOA), including those who are at increased risk (AIR) of respiratory syncytial virus (RSV)-lower respiratory tract disease (LRTD), versus adults >=60 YOA

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.

  1. Specific inclusion criteria for all participants in Cohort 1 (Adults HA-RSV Group, Adults HA-Placebo Group, Adults AIR-RSV Group & Adults AIR-Placebo Group)
* A male or female participant 50-59 YOA at the time of the study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception from 1 month prior to study intervention administration until study end for this study, and
  * has a negative pregnancy test on the day of study intervention administration.

Specific inclusion criteria for participants in the Adults-HA Sub-cohort

* Healthy participants as established by medical history and clinical examination before entering into the study.
* Participants with chronic stable medical conditions with or without specific treatment, such as hypertension, hypercholesterolemia, or hypothyroidism, and who are not at increased risk for RSV-LRTD , are allowed to participate in this study if considered by the investigator as medically stable (no changes in the treatment or disease severity in the past 3 months).

Specific inclusion criteria for participants in the Adults-AIR Sub cohort

Participants should be diagnosed with at least 1 of the following medical conditions and have a stable condition (no changes in the treatment or disease severity in the past 3 months):

* Chronic pulmonary disease resulting in activity restricting symptoms or use of long-term medication
* Chronic cardiovascular disease
* Diabetes mellitus: types 1 and 2
* Other diseases at increased risk for RSV-LRTD disease

  * Chronic kidney disease
  * Chronic liver disease 2. Specific inclusion criteria for Cohort 2 (OA-RSV Group)
* A male or female participant ≥60 YOA at the time of the study intervention administration.
* Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease are allowed to participate in this study if considered by the investigator as medically stable (no changes in the treatment or disease severity in the past 3 months).
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Hypersensitivity to latex.
* Unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol. Study participants may decide to assign a caregiver to help them complete the study procedures.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study intervention during the period beginning 30 days before the dose of study intervention (Day -29 to Day 1), or planned use during the study period (up to Visit 4, Month 12).
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of study intervention administration, with the exception of inactivated and subunit influenza vaccines or COVID-19 vaccines (fully licensed or with EUA) which can be administered up to 14 days before or from 14 days after the study intervention administration.

Note: In case an emergency mass vaccination for an unforeseen public health threat is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.

* Previous vaccination with an RSV vaccine, including investigational RSV vaccines.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or administration of long-acting immune modifying treatments or planned administration at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration:
  * For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
  * Administration of immunoglobulins and/or any blood products or plasma derivatives.
  * Up to 6 months prior to study intervention administration: long-acting immune modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or invasive medical device).

Other exclusions Other exclusions for all participants

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study period that will prohibit participating in the study until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.

Other exclusions for Cohort 1

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1544 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2024-02-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Ferguson M, Schwarz TF, Nunez SA, Rodriguez-Garcia J, Mital M, Zala C, Pek B, Schmitt B, Toursarkissian N, Ochoa Mazarro D, Grosskopf J, Voors-Pette C, Mehta H, Amare Hailemariam H, Gerard C, Damaso S, David MP, Descamps D, Hill J, Vandermeulen C, Hulstrom V. Immune persistence and safety of the AS01E-adjuvanted respiratory syncytial virus prefusion F protein-based vaccine in adults 50-59 years of age, including at-increased-risk adults: A randomized controlled trial. Hum Vaccin Immunother. 2025 Dec;21(1):2579335. doi: 10.1080/21645515.2025.2579335. Epub 2025 Nov 5. PMID 41194599
- [Derived] Ferguson M, Schwarz TF, Nunez SA, Rodriguez-Garcia J, Mital M, Zala C, Schmitt B, Toursarkissian N, Mazarro DO, Grosskopf J, Voors-Pette C, Mehta H, Hailemariam HA, de Heusch M, Salaun B, Damaso S, David MP, Descamps D, Hill J, Vandermeulen C, Hulstrom V; RSV OA=ADJ-018 Study Group. Noninferior Immunogenicity and Consistent Safety of Respiratory Syncytial Virus Prefusion F Protein Vaccine in Adults 50-59 Years Compared to >/=60 Years of Age. Clin Infect Dis. 2024 Oct 15;79(4):1074-1084. doi: 10.1093/cid/ciae364. PMID 39099093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 1544 participants enrolled in this study, 1534 participants received at least one study intervention, from which 1 participant in OA-RSV group received placebo instead of RSVPreF3 OA vaccine and was excluded from the group. Therefore, the Exposed set included 1533 participants.
Period: Overall Study
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Started | 383 | 192 | 386 | 191 | 381
Completed | 363 | 184 | 369 | 180 | 369
Not Completed | 20 | 8 | 17 | 11 | 12
Not completed — Lost to Follow-up | 13 | 1 | 7 | 3 | 4
Not completed — Consent withdrawal, not due to a (S)AE | 4 | 6 | 4 | 2 | 7
Not completed — Other | 2 | 0 | 2 | 2 | 0
Not completed — Migrated / moved from the study area | 1 | 1 | 0 | 3 | 1
Not completed — Adverse event requiring expedited reporting | 0 | 0 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adults HA-RSV Group: Healthy adults or adults with chronic stable conditions with or without treatment that do not lead to an increased risk of RSV-LRTD, aged 50-59 years old received 1 dose of RSVPreF3 OA vaccine at Day 1 and were followed until study end.
- Total: Total of all reporting groups
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group | Total
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381 | 1533
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 54.8 (2.8) | 54.7 (2.8) | 55.3 (2.8) | 55.6 (2.8) | 64.1 (2.9) | 58.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 119 | 186 | 85 | 188 | 799
  Male | 162 | 73 | 200 | 106 | 193 | 734
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 23 | 63 | 35 | 50 | 219
  Not Hispanic or Latino | 335 | 168 | 323 | 156 | 330 | 1312
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: RSV-A Neutralization Titers Expressed as Group Geometric Mean Titer (GMT) in Healthy Participants Compared to OA-RSV Group
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were expressed in Estimated Dilution 60 (ED60) and were measured on blood samples collected from vaccinated subjects. The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing antibodies included the baseline value as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included Adult HA-RSV and OA-RSV groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At 1 month after the RSVPreF3 OA vaccine administration (Day 31)
Population: Analysis was performed on the per protocol set (PPS) for humoral analysis which included all eligible participants who received the study intervention as per protocol, had RSV-A immunogenicity results pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on the administered intervention.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | OA-RSV Group
Number analyzed (Participants) | 326 | 343
Titer | 7906.0 [7178.1 to 8707.7] | 7518.9 [6843.2 to 8261.3]
Statistical Analysis 1: Comparison: Adults HA-RSV Group vs OA-RSV Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when administered to healthy adults aged 50-59 years of age compared with older adults aged 60 years of age or above; Test type: Non-Inferiority — Non-inferiority is demonstrated if the anti-RSV-A GMT ratio (OA-RSV Group over Adults-HA-RSV Group) is less than (<) 1.5 at 1 month post RSVPreF3 OA vaccine administration; GMT Ratio = 0.95, 95% CI 2-sided [0.83 to 1.09] — The comparison is done using the group ratio of adjusted GMT (OA-RSV/Adults-HA-RSV) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate

2. Primary Outcome: RSV-A Neutralization Titers Expressed as Group Seroresponse Rate (SRR) Difference in Healthy Participants Compared to OA-RSV Group
Description: The SRR is defined as the proportion of participants having a fold increase in neutralization titers (1 month post-study intervention administration over pre-study intervention administration) greater than or equal to 4 (>=4).
Time Frame: At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31) compared to baseline (Day 1)
Population: Analysis was performed on PPS for humoral analysis which included all eligible participants who received the study intervention as per protocol, had SRR results for RSV-A at pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on the administered intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | OA-RSV Group
Number analyzed (Participants) | 270 | 275
Percentage of participants | 82.8 [78.3 to 86.8] | 80.2 [75.6 to 84.3]
Statistical Analysis 1: Comparison: Adults HA-RSV Group vs OA-RSV Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI on the group difference (OA-RSV Group minus Adults-HA-RSV Group) in terms of SRR is <10%, at 1 month post RSVPreF3 OA vaccine administration; Difference in percentage = -2.65, 95% CI 2-sided [-8.54 to 3.28] — The comparison is done using the difference of SRR (OA-RSV -Adults-HA-RSV)

3. Primary Outcome: RSV-B Neutralization Titers Expressed as Group GMT in Healthy Participants Compared to OA-RSV Group
Description: Serological assays for the determination of antibodies against RSV-B were performed by neutralization assay. The corresponding antibody titers were expressed in ED60. The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing antibodies included the baseline value as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included Adult HA-RSV and OA-RSV groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At 1 month after the RSVPreF3 OA vaccine administration (Day 31)
Population: Analysis was performed on PPS for humoral analysis which included all eligible participants who received the study intervention as per protocol, had RSV-B immunogenicity results pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on the administered intervention.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | OA-RSV Group
Number analyzed (Participants) | 326 | 342
Titer | 9024.8 [8240.8 to 9883.3] | 8070.3 [7385.2 to 8819.1]
Statistical Analysis 1: Comparison: Adults HA-RSV Group vs OA-RSV Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority is demonstrated if the anti-RSV-B GMT ratio (OA-RSV Group over Adults-HA-RSV Group) is <1.5 at 1 month post RSVPreF3 OA vaccine administration; GMT Ratio = 0.89, 95% CI 2-sided [0.79 to 1.02] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: RSV-B Neutralization Titers Expressed as Group SRR in Healthy Participants Compared to OA-RSV Group
Description: The SRR is defined as the proportion of participants having a fold increase in neutralization titers (1 month post-study intervention administration over pre-study intervention administration) >=4.
Time Frame: At 1 month after the RSVPreF3 OA vaccine administration (Day 31) compared to baseline (Day 1)
Population: Analysis was performed on PPS for humoral analysis which included all eligible participants who received the study intervention as per protocol, had SRR results for RSV-B at pre- and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Analysis per group is based on the administered intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | OA-RSV Group
Number analyzed (Participants) | 255 | 254
Percentage of participants | 78.2 [73.3 to 82.6] | 74.3 [69.3 to 78.8]
Statistical Analysis 1: Comparison: Adults HA-RSV Group vs OA-RSV Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -3.95, 95% CI 2-sided [-10.39 to 2.53] — The comparison is done using the difference of SRR (OA-RSV -Adults-HA-RSV)

5. Primary Outcome: RSV-A Neutralization Titers Expressed as Group GMT Titer in Participants at Increased Risk of RSV-LRTD (Adults-AIR-RSV Group) Compared to OA-RSV Group
Description: Serological assays for the determination of antibodies against RSV-A are performed by neutralization assay. The corresponding antibody titers were expressed in ED60. The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing antibodies included the baseline value as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included Adult AIR-RSV and OA-RSV groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults AIR-RSV Group | OA-RSV Group
Number analyzed (Participants) | 342 | 343
Titer | 8925.1 [8117.9 to 9812.6] | 7460.7 [6786.8 to 8201.5]
Statistical Analysis 1: Comparison: Adults AIR-RSV Group vs OA-RSV Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when administered to adults at increased risk of RSV-LRTD aged 50-59 years of age compared with older adults aged 60 years of age or above; Test type: Non-Inferiority — Non-inferiority is demonstrated if the anti-RSV-A GMT ratio (OA-RSV Group over Adults-AIR-RSV Group) is <1.5 at 1 month post RSVPreF3 OA vaccine administration; GMT Ratio = 0.84, 95% CI 2-sided [0.73 to 0.96] — The comparison is done using the group ratio of adjusted GMT (OA-RSV/Adults-AIR-RSV) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate

6. Primary Outcome: RSV-A Neutralization Titers Expressed as Group SRR in Participants at Increased Risk of RSV-LRTD (Adults-AIR-RSV Group) Compared to OA-RSV Group
Description: as for outcome 4
Time Frame: At 1 month after the RSVPreF3 OA vaccine administration (Day 31) compared to baseline (Day 1)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults AIR-RSV Group | OA-RSV Group
Number analyzed (Participants) | 297 | 275
Percentage of participants | 86.8 [82.8 to 90.2] | 80.2 [75.6 to 84.3]
Statistical Analysis 1: Comparison: Adults AIR-RSV Group vs OA-RSV Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI on the group difference (OA-RSV Group over Adults-AIR-RSV Group) in terms of SRR is <10%, at 1 month post RSVPreF3 OA vaccine administration; Difference in percentage = -6.67, 95% CI 2-sided [-12.26 to -1.12] — The comparison is done using the difference of SRR (OA-RSV -Adults-AIR-RSV)

7. Primary Outcome: RSV-B Neutralization Titers Expressed as Group GMT in Participants at Increased Risk of RSV-LRTD (Adults-AIR-RSV Group) Compared to OA-RSV Group
Description: Serological assays for the determination of antibodies against RSV-B are performed by neutralization assay. The corresponding antibody titers were expressed in ED60. The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing antibodies included the baseline value as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included Adult AIR-RSV and OA-RSV groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At 1 month after the RSVPreF3 OA vaccine administration (Day 31)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults AIR-RSV Group | OA-RSV Group
Number analyzed (Participants) | 342 | 342
Titer | 10048.6 [9218.4 to 10953.5] | 8073.4 [7406.4 to 8800.4]
Statistical Analysis 1: Comparison: Adults AIR-RSV Group vs OA-RSV Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — Non-inferiority is demonstrated if the anti-RSV-B GMT ratio (OA-RSV Group over Adults-AIR-RSV Group) is <1.5 at 1 month post RSVPreF3 OA vaccine administration; GMT Ratio = 0.80, 95% CI 2-sided [0.71 to 0.91] — [estimate comment as in outcome 5, analysis 1]

8. Primary Outcome: RSV-B Neutralization Titers Expressed as Group SRR in Participants at Increased Risk of RSV-LRTD (Adults-AIR-RSV Group) Compared to OA-RSV Group
Description: as for outcome 4
Time Frame: At 1 month after the RSVPreF3 OA investigational vaccine administration (Day 31) compared to baseline (Day 1)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults AIR-RSV Group | OA-RSV Group
Number analyzed (Participants) | 279 | 254
Percentage of participants | 81.6 [77.1 to 85.5] | 74.3 [69.3 to 78.8]
Statistical Analysis 1: Comparison: Adults AIR-RSV Group vs OA-RSV Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage = -7.31, 95% CI 2-sided [-13.52 to -1.09] — The comparison is done using the difference of SRR (OA-RSV -Adults-AIR-RSV)

9. Secondary Outcome: Percentage of Participants Reporting Each Solicited Administration Site Event (Pain, Redness and Swelling)
Description: Assessed solicited administration site events were pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Any erythema and swelling symptom = symptom reported with a surface diameter greater than 0 millimeters.
Time Frame: During the 4-day follow up period after vaccination (vaccine or placebo administered on Day 1)
Population: Analysis was based on the Exposed Set (ES), which included all participants who received the study intervention and had data for solicited administration site events analysis at the assessed timeframe.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 377 | 191 | 379 | 189 | 379
Percentage of participants
  Erythema | 11.9 [8.8 to 15.6] | 0.5 [0.0 to 2.9] | 14.5 [11.1 to 18.5] | 0.5 [0.0 to 2.9] | 12.1 [9.0 to 15.9]
  Pain | 76.7 [72.1 to 80.8] | 10.5 [6.5 to 15.7] | 75.2 [70.5 to 79.5] | 14.3 [9.6 to 20.1] | 61.2 [56.1 to 66.1]
  Swelling | 9.3 [6.6 to 12.7] | 1.0 [0.1 to 3.7] | 11.6 [8.6 to 15.3] | 0.5 [0.0 to 2.9] | 7.7 [5.2 to 10.8]

10. Secondary Outcome: Percentage of Participants Reporting Each Solicited Systemic Event (Fever, Headache, Muscle Pain, Joint Pain, Tiredness)
Description: Assessed solicited systemic events were arthralgia, fatigue, headache, myalgia and fever [temperature equal to or above (>=) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relation to study intervention.
Time Frame: During the 4-day follow up period after vaccination (vaccine or placebo administered on Day 1)
Population: Analysis was based on the Exposed Set (ES), which included all participants who received the study intervention and had data for solicited systemic events analysis at the assessed timeframe.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 377 | 191 | 379 | 190 | 379
Percentage of participants
  Arthralgia | 26.0 [21.6 to 30.7] | 5.8 [2.9 to 10.1] | 20.8 [16.9 to 25.3] | 10.0 [6.1 to 15.2] | 12.9 [9.7 to 16.7]
  Fatigue | 44.0 [39.0 to 49.2] | 17.3 [12.2 to 23.4] | 36.1 [31.3 to 41.2] | 19.5 [14.1 to 25.8] | 24.0 [19.8 to 28.6]
  Headache | 35.8 [31.0 to 40.9] | 16.8 [11.8 to 22.8] | 27.7 [23.3 to 32.5] | 17.4 [12.3 to 23.5] | 21.1 [17.1 to 25.6]
  Myalgia | 39.3 [34.3 to 44.4] | 5.8 [2.9 to 10.1] | 32.5 [27.8 to 37.4] | 14.2 [9.6 to 20.0] | 21.4 [17.4 to 25.8]
  Fever | 3.7 [2.0 to 6.2] | 1.0 [0.1 to 3.7] | 2.6 [1.3 to 4.8] | 1.1 [0.1 to 3.8] | 1.6 [0.6 to 3.4]

11. Secondary Outcome: Percentage of Participants Reporting Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs are defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: During the 30-day follow up period after vaccination (vaccine or placebo administered on Day 1)
Population: Analysis was based on the Exposed Set (ES), which included all participants who received the study intervention and had data for assessed timeframe and unsolicited events analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 13.6 [10.3 to 17.4] | 13.5 [9.0 to 19.2] | 15.3 [11.8 to 19.3] | 10.5 [6.5 to 15.7] | 16.3 [12.7 to 20.4]

12. Secondary Outcome: Percentage of Participants Reporting Any Serious Adverse Events (SAEs) Within 6 Months of Vaccination
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, or results in an abnormal pregnancy outcome.
Time Frame: From the day of the vaccination up to 6 months after vaccination (vaccine or placebo administered on Day 1)
Population: Analysis was based on the ES, which included all participants who received the study intervention. Analysis per group is based on the administered intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 0.8 [0.2 to 2.3] | 2.1 [0.6 to 5.2] | 3.9 [2.2 to 6.3] | 2.1 [0.6 to 5.3] | 2.4 [1.1 to 4.4]

13. Secondary Outcome: Percentage of Participants Reporting Any Onset Potential Immune Mediated Diseases (pIMDs) Within 6 Months of Vaccination
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From the day of the vaccination up to 6 months after vaccination (vaccine or placebo administered on Day 1)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 0 [0 to 1.0] | 0 [0 to 1.9] | 1.0 [0.3 to 2.6] | 0.5 [0.0 to 2.9] | 0.8 [0.2 to 2.3]

14. Secondary Outcome: Percentage of Participants Reporting SAEs Related to Study Intervention Administration Within 12 Months of Vaccination
Description: as for outcome 12
Time Frame: From the day of the vaccination up to 12 months after vaccination (vaccine or placebo administered on Day 1)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 0 [0 to 1.0] | 0 [0 to 1.9] | 0 [0 to 1.0] | 0 [0.0 to 1.9] | 0.3 [0.0 to 1.5]

15. Secondary Outcome: Percentage of Participants Reporting pIMDs Related to Study Intervention Administration Within 12 Months of Vaccination
Description: as for outcome 13
Time Frame: From the day of the vaccination up to 12 months after vaccination (vaccine or placebo administered on Day 1)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 0 [0 to 1.0] | 0 [0 to 1.9] | 0 [0 to 1.0] | 0 [0.0 to 1.9] | 0.3 [0.0 to 1.5]

16. Secondary Outcome: Percentage of Participants Reporting Any Fatal SAEs
Description: as for outcome 12
Time Frame: From the day of the vaccination up to 12 months after vaccination (vaccine or placebo administered on Day 1)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 383 | 192 | 386 | 191 | 381
Percentage of participants | 0 [0 to 1.0] | 0 [0 to 1.9] | 1.0 [0.3 to 2.6] | 0.5 [0.0 to 2.9] | 0 [0 to 1.0]

17. Secondary Outcome: RSV-A Neutralization Titers Expressed as GMT, up to One Month Post-intervention
Description: Serological assays for the determination of antibodies against RSV-A are performed by neutralization assay. The corresponding antibody titers were expressed in ED60. Unadjusted GMTs were provided for Adult HA-RSV, Adults HA-Placebo, Adult AIR-RSV, Adult AIR-Placebo and OA-RSV groups.
Time Frame: At pre-study intervention administration (Day 1) and 1 month after study intervention administration (Day 31)
Population: Analysis was performed on PPS for humoral analysis which included all eligible participants who received the study intervention as per protocol, had immunogenicity results pre- and post-dose for the assessed analysis, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only those participants with data available at the time of the analysis were reported in this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 347 | 181 | 364 | 186 | 364
Titer
  Day 1 | 768.8 [704.7 to 838.9] | 772.0 [677.9 to 879.1] | 779.5 [725.5 to 837.6] | 729.8 [648.6 to 821.0] | 775.7 [709.9 to 847.5]
  Day 31: number analyzed (Participants) | 329 | 177 | 344 | 178 | 348
  Day 31 | 7925.4 [7125.6 to 8815.0] | 796.9 [696.4 to 912.0] | 8804.1 [7953.3 to 9746.0] | 774.7 [683.0 to 878.6] | 7498.8 [6759.5 to 8319.1]

18. Secondary Outcome: RSV-A Neutralization Titers Expressed as GMT at Month 6 and Month 12 Post-intervention
Description: as for outcome 17
Time Frame: At 6 months and at 12 months after study intervention administration
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 317 | 171 | 345 | 178 | 355
Titer
  Month 6 | 3850.7 [3448.6 to 4299.7] | 849.6 [748.9 to 963.9] | 3980.6 [3608.6 to 4391.1] | 854.2 [756.2 to 965.0] | 3846.3 [3469.7 to 4263.7]
  Month 12: number analyzed (Participants) | 306 | 166 | 327 | 170 | 334
  Month 12 | 3192.9 [2855.1 to 3570.7] | 965.1 [846.8 to 1099.9] | 3075.1 [2772.2 to 3411.0] | 971.8 [864.6 to 1092.4] | 3080.4 [2764.8 to 3432.0]

19. Secondary Outcome: RSV-B Neutralization Titers Expressed as GMT, up to One Month Post-intervention
Description: Serological assays for the determination of antibodies against RSV-B are performed by neutralization assay. The corresponding antibody titers were expressed in ED60. Unadjusted GMTs were provided for Adult HA-RSV, Adults HA-Placebo, Adult AIR-RSV, Adult AIR-Placebo and OA-RSV groups.
Time Frame: At pre-study intervention administration (Day 1) and 1 month after study intervention administration (Day 31)
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 347 | 181 | 364 | 186 | 364
Titer
  Day 1 | 1091.1 [1000.3 to 1190.2] | 1197.7 [1055.7 to 1358.8] | 1141.4 [1050.5 to 1240.0] | 1167.2 [1035.0 to 1316.1] | 1109.1 [1020.6 to 1205.3]
  Day 31: number analyzed (Participants) | 329 | 177 | 344 | 178 | 347
  Day 31 | 8971.9 [8109.6 to 9925.8] | 1145.3 [1012.4 to 1295.5] | 9943.0 [9035.8 to 10941.4] | 1141.8 [1007.4 to 1294.2] | 8169.3 [7412.6 to 9003.3]

20. Secondary Outcome: RSV-B Neutralization Titers Expressed as GMT, at Month 6 and Month 12 Post-intervention
Description: as for outcome 19
Time Frame: At 6 months and at 12 months after study intervention administration
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 317 | 171 | 345 | 178 | 355
Titer
  Month 6 | 3880.7 [3488.4 to 4317.0] | 1003.2 [875.5 to 1149.4] | 4020.8 [3635.9 to 4446.5] | 942.1 [825.4 to 1075.3] | 3710.4 [3361.0 to 4096.1]
  Month 12: number analyzed (Participants) | 306 | 166 | 327 | 170 | 334
  Month 12 | 3562.8 [3176.0 to 3996.7] | 1218.6 [1038.8 to 1429.5] | 3669.9 [3287.1 to 4097.3] | 1153.5 [996.6 to 1335.2] | 3527.7 [3177.5 to 3916.4]

21. Secondary Outcome: Frequency of RSVPreF3-specific Cluster of Differentiation (CD)4+ T Cells Expressing at Least 2 Activation Markers up to One Month Post-intervention
Description: Among markers expressed are interleukin-2/13/17 (IL-2, IL-13, IL-17), cluster of 40 ligand (CD40L), 41BB, tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At pre-study intervention administration (Day 1) and 1 month after study intervention administration (Day 31)
Population: Analysis was performed on Cell-Mediated immune (CMI) sub-cohort of the PPS,which included all eligible participants who received the study intervention as per protocol,had immunogenicity results pre- and post-dose for RSVPreF3 OA specific CD4+T cells, complied with blood draw intervals,without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.Only the participants with data available at the time of the analysis were reported
Measure: Geometric Mean (Standard Deviation); unit: CD4+ T cells/million cells
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 47 | 28 | 55 | 27 | 26
CD4+ T cells/million cells
  Day 1: number analyzed (Participants) | 47 | 28 | 55 | 23 | 26
  Day 1 | 102.7 (0.9) | 125.6 (0.9) | 161.5 (0.6) | 114.7 (0.9) | 111.3 (0.9)
  Day 31: number analyzed (Participants) | 45 | 27 | 46 | 27 | 24
  Day 31 | 1282.5 (0.4) | 167.7 (0.8) | 1043.6 (0.6) | 131.9 (0.8) | 1016.9 (0.8)

22. Secondary Outcome: Frequency of RSVPreF3-specific CD4+ T Cells Expressing at Least 2 Activation Markers, at Month 6 and Month 12 Post-intervention
Description: as for outcome 21
Time Frame: At 6 months and at 12 months after study intervention administration
Population: Analysis was performed on CMI sub-cohort of the PPS, which included all eligible participants who received the study intervention as per protocol, had immunogenicity results pre- and post-dose for RSVPreF3 OA specific CD4+ T cells, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only the participants with data available at the time of the analysis were reported.
Measure: Geometric Mean (Standard Deviation); unit: CD4+ T cells/million cells
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 58 | 36 | 56 | 27 | 31
CD4+ T cells/million cells
  Month 6: number analyzed (Participants) | 52 | 28 | 55 | 26 | 28
  Month 6 | 825.6 (0.3) | 140.5 (0.8) | 662.9 (0.3) | 39.2 (1.0) | 763.5 (0.5)
  Month 12 | 492.0 (0.6) | 175.8 (0.5) | 335.5 (0.7) | 59.4 (1.0) | 414.1 (0.7)

23. Secondary Outcome: Frequency of RSVPreF3-specific CD8+ T Cells Expressing at Least 2 Activation Markers, up to One Month Post-intervention
Description: Among markers expressed are IL-2, IL-13, IL-17, CD40L, 41BB, TNF-α and IFN-γ, in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At pre-study intervention administration (Day 1) and 1 month after study intervention administration (Day 31)
Population: Analysis was performed on CMI sub-cohort of the PPS, which included all eligible participants who received the study intervention as per protocol, had immunogenicity results pre- and post-dose for RSVPreF3 OA specific CD8+ T cells, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only the participants with data available at the time of the analysis were reported.
Measure: Geometric Mean (Standard Deviation); unit: CD8+ T cells/million cells
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 46 | 28 | 55 | 27 | 26
CD8+ T cells/million cells
  Day 1: number analyzed (Participants) | 46 | 28 | 55 | 23 | 26
  Day 1 | 10.1 (1.1) | 6.0 (0.9) | 15.5 (1.0) | 10.8 (1.1) | 12.0 (1.0)
  Day 31: number analyzed (Participants) | 45 | 27 | 46 | 27 | 24
  Day 31 | 15.2 (1.1) | 11.9 (1.1) | 18.1 (1.1) | 4.8 (1.1) | 12.0 (1.2)

24. Secondary Outcome: Frequency of RSVPreF3-specific CD8+ T Cells Expressing at Least 2 Activation Markers, at Month 6 and Month 12
Description: as for outcome 23
Time Frame: At 6 months and at 12 months after study intervention administration
Population: as for outcome 23
Measure: Geometric Mean (Standard Deviation); unit: CD8+ T cells/million cells
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
Number analyzed (Participants) | 58 | 36 | 56 | 27 | 31
CD8+ T cells/million cells
  Month 6: number analyzed (Participants) | 52 | 28 | 55 | 26 | 28
  Month 6 | 23.1 (1.0) | 12.2 (1.1) | 27.6 (1.0) | 14.0 (1.0) | 14.8 (1.1)
  Month 12 | 15.2 (1.0) | 23.0 (0.9) | 16.2 (1.0) | 6.6 (1.1) | 14.9 (1.0)

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 (day of vaccination) up to Day 4 post-dose. Unsolicited AEs were collected from Day 1 up to Day 30 post-dose. SAEs and pIMDs were collected from Day 1 up to Month 6 post dose-administration. Related SAEs, related pIMDs and fatal SAEs were collected from Day 1 up to study end (Month 12).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Adults HA-RSV Group | Adults HA-Placebo Group | Adults AIR-RSV Group | Adults AIR-Placebo Group | OA-RSV Group
All-Cause Mortality (participants affected / at risk) | 0/383 | 0/192 | 1/386 | 1/191 | 0/381
Serious Adverse Events (participants affected / at risk) | 3/383 | 4/192 | 15/386 | 4/191 | 9/381
Other Adverse Events (participants affected / at risk) | 325/383 | 76/192 | 318/386 | 74/191 | 279/381
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults HA-RSV Group (N=383) | Adults HA-Placebo Group (N=192) | Adults AIR-RSV Group (N=386) | Adults AIR-Placebo Group (N=191) | OA-RSV Group (N=381)
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kyphosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults HA-RSV Group (N=383) | Adults HA-Placebo Group (N=192) | Adults AIR-RSV Group (N=386) | Adults AIR-Placebo Group (N=191) | OA-RSV Group (N=381)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular retrobulbar haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor dental condition (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Administration site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 166 (167) | 34 (34) | 136 (136) | 37 (37) | 92 (92)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 40 (40) | 1 (1) | 55 (55) | 1 (1) | 42 (42)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 32 (32) | 2 (2) | 43 (43) | 1 (1) | 25 (25)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 14 (14) | 2 (2) | 11 (11) | 3 (3) | 7 (7)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 7 (7) | 0 (0) | 5 (5)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 101 (102) | 12 (12) | 80 (81) | 19 (19) | 50 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 149 (150) | 12 (13) | 123 (123) | 27 (27) | 83 (84)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 137 (139) | 34 (35) | 106 (106) | 33 (34) | 81 (81)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 289 (289) | 20 (20) | 285 (285) | 27 (27) | 232 (232)
Administration site erythema (General disorders) | 40 (40) | 1 (1) | 55 (55) | 1 (1) | 42 (42)
Administration site swelling (General disorders) | 32 (32) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT05590403/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT05590403/SAP_002.pdf